CLINICAL TRIAL: NCT03643172
Title: Termination of Nucleos(t)Ide Analogue Therapy of HBeAg Negative Chronic Hepatitis B - 2nd Register Study
Brief Title: Terminator 2 Register
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: German Center for Infection Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2018-06-19; First posted 2018-08-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-08

CONDITIONS: Chronic Hepatitis B, HBeAg Negative
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients with chronic HBeAg negative hepatitis B treated with nucleos(t)ide analogues, who discontinue treatment based in the criteria outlined in the EASL hepatitis B guidelines shall be included in the present study. The aim is to evaluate the clinical outcome (virological relapse, HBsAg decline) and associated virological and immunological parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with chronic hepatitis B virus infection documented by detectable HBsAg.
2. Age > 18 years
3. Ongoing antiviral therapy with Entecavir or Tenofovir (TDF)
4. At least 3 years HBV-DNA < 20 IU/ml (=100 copies/ml)
5. HBeAg negative
6. Willingness to give written informed consent and willingness to participate and to comply with the protocol.

Exclusion Criteria:

1. HIV infection, persistent HDV-infection, persistent HCV infection
2. History or other evidence of a medical condition associated with chronic liver disease other than HBV associated (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures).
3. History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
4. Patients with advanced liver fibrosis and liver cirrhosis (fibroscan >10.0 kPa)
5. Patients with hepatocellular carcinoma
6. History of major organ transplantation or other immunosuppressive conditions
7. History or other evidence of severe illness, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
8. History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 12 months prior to cessation of antiviral therapy or the expectation that such treatment will be needed at any time during the study

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Non-cirrhotic male and female patients with chronic hepatitis B virus infection documented by detectable HBsAg.
  2. Age > 18 years
  3. ongoing antiviral therapy with Entecavir or Tenofovir (TDF)
  4. At least 3 years HBV-DNA < 20 IU/ml (=100 copies/ml)
  5. HBeAg negative
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
HBsAg | 48 weeks
  HBsAg Change > 1 log 48 weeks after stopping NA

SECONDARY OUTCOMES:
Virological relapse | at every visit up to 96 weeks
  HBV DNA > 2,000 IU/ml
Biochemical relapse | at every visit up to 96 weeks
  ALT > 2 x upper limit of normal
Retreatment | at every visit up to 48 weeks
  Retreatment until week 48 according to current EASL guidelines
Negativity for HBsAg | at every visit up to 96 weeks
  HBsAg negative until week 96 of follow-up
timepoint of relapse | at every visit up to 96 weeks
  timepoint of relapse
T cell response | at every visit up to 96 weeks
  > 3x change of T cell responses from baseline after in vitro culture with HBV specific peptides
Cytokine response | at every visit up to 96 weeks
  > 3x change of cytokines from baseline measured by ELISA and Multiplex assay
Chance in HBcrAg | at every visit up to 96 weeks
  Chance in HBcrAg (U/mL)
Change in HBV RNA | at every visit up to 96 weeks
  Chance in HBV RNA (U/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohlendorf V, Wubbolding M, Honer Zu Siederdissen C, Bremer B, Deterding K, Wedemeyer H, Cornberg M, Maasoumy B. Limited Value of HBV-RNA for Relapse Prediction After Nucleos(t)ide Analogue Withdrawal in HBeAg-negative Hepatitis B Patients. J Viral Hepat. 2025 Apr;32(4):e14026. doi: 10.1111/jvh.14026. Epub 2024 Oct 19. PMID 39425534